CLINICAL TRIAL: NCT03569722
Title: EpxCogScreen -- A Phone-based Rapid Cognitive Screen (RCS)
Status: Terminated | Type: Observational
Why Stopped: This study was terminated due to insufficient recruitment.
Sponsor: Theodore Malmstrom, PhD (Other)
Responsible Party: Sponsor-Investigator, Theodore Malmstrom, PhD, Primary Investigator, St. Louis University
Organization: St. Louis University (Other)
Other Study IDs: 27943
Record Dates: First submitted 2018-05-11; First posted 2018-06-26 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Dementia; Telemedicine; Cognitive Dysfunction
Keywords: Cognitive screen
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults: Older adults, ages 65+

SUMMARY:
EpxCogScreen is a phone-based intervention to administer the Rapid Cognitive Screen, a validated screening tool for dementia, over SMS text messaging. The results of the screen are sent to the physician automatically, which allows physicians to monitor their patients and gives them the ability to respond rapidly to any concerns of cognitive decline. In this study, patients' at-home RCS scores done by EpxCogScreen will be compared to their in-clinic RCS scores, and to clinical diagnosis of dementia (where available), to investigate the validity of EpxCogScreen.

DETAILED DESCRIPTION:
Telemedicine is a modern field of clinical medicine that incorporates telecommunication and information technology to diagnose and manage health care remotely. Interventions range from telephone reminders to remote physician consultation by video conference. Simple technology such as telephones and SMS texting are ubiquitous forms of communication that have the potential to increase the frequency of physician-patient contact. Use of SMS messaging, for example, may help to improve patient adherence, promote education and engagement, allow real-time collection of critical biometric and clinical data over time, and bridge the gap between recognizing adverse events and actual disease management.

One geriatric syndrome that may benefit from early detection is dementia. Dementia is characterized by impairments in cognitive function, such as memory, comprehension, visual-spatial orientation, language, and/or judgement. The most common form of dementia is Alzheimer's disease, but vascular dementia and Lewy-body dementia can also cause cognitive impairment. It is estimated that 47.5 million people are affected with dementia worldwide and it is the most common form of disability in the geriatric population over the age of 65, affecting 1 in 9 people in that population [van der Linde, et al., 2016]. A formal diagnosis for Alzheimer's relies primarily on clinical evaluation by a clinician (e.g., neurologist, psychiatrist), usually in conjunction with results from neuropsychological testing and/or informant reports re patients' memory and thinking.

In 2011, the Affordable Care Act added routine cognitive screening as a component of the Medicare Annual Wellness Visit, but did not recommend a universal screening tool [Cordell et al., 2012]. This initiative was supported by many public organizations, including the Alzheimer's Association. The U.S. Preventative Services Task Force (USPSTF) currently does not recommend universal cognitive screening for older adults [Lin et al., 2013]. Nonetheless, there may be benefits to case finding among older adults patients through the use of screening measures. For example, early intervention has been shown to delay placement into nursing homes, empower patients to be more involved with their care plan, and allow physicians to identify and manage comorbidities such as depression, malnutrition, and falls more effectively [Dubois et al., 2016; Weimer et al., 2009]. Delayed admission into nursing homes and fewer hospitalizations are associated with decreased healthcare costs for patients, their families, and the healthcare system [Weimer et al., 2009]. It also has been reported that a lot of Alzheimer's patients are undiagnosed, in part, because screening has not yet reached standard-of-practice in geriatric and primary care clinics [Dubois et al., 2016].

Healthcare professionals may not be able to regularly screen for cognitive dysfunction due to time constraints in clinical practice. Typical neuropsychological tests for cognitive dysfunction, such as the Mini-Mental State Exam (MMSE), are administered in the physician's office and can take 7 to 15 minutes to complete. The Rapid Cognitive Screen (RCS) is a 3-item screening tool that takes less than 5 minutes to complete. This screen has exhibited good sensitivity and specificity in detecting both mild cognitive impairment and dementia in patients over the age of 65 [Malmstrom et al., 2015]. EpxCogScreen utilizes the RCS to create a phone-based screen for cognitive dysfunction that can be done in-home when administered by a caregiver.

In this study, the RCS will be administered in a healthcare clinic using standard procedures, and at home using a telemedicine (text-based) format called EpxCogScreen. Patients-caregiver dyads will be recruited from a geriatric medicine clinic at an academic medical health center. A healthcare professional will administer the RCS to a patient in the clinic, one month subsequent to this, a caregiver will administer the RCS to patients in-home via EpxCogScreen using SMS messaging on a smartphone. Each caregiver will be given the option to receive RCS administration instructions via text, or to use directions from a handout that the caregiver received while in clinic. Patient responses will be recorded through text. Physicians will be notified immediately through EpxCogScreen system if a patients in-home RCS score is 3 or more points lower than their RCS score from the previous month's healthcare clinic visit. Individuals will have the ability to opt out of the study electronically via text and phone at any point during the study.

The association of in-home RCS scores with the clinic RCS scores and with the clinical diagnosis of cognitive dysfunction in medical records will be investigated in this study. Data analysis will evaluate the association of RCS components (recall, clock drawing, insight) and total scores for in-home versus clinic measurements; and the sensitivity and specificity of the in-home, SMS text-based RCS will be determined by comparison to clinical diagnosis of cognitive dysfunction from chart review, and by comparison to RCS clinic results.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >65 years old
* Patients must have a caregiver or family member who can administer the intervention at home
* Caregivers must be between 18-90 years old
* Caregivers must have a working cellular device with SMS texting capabilities
* Both patients and caregivers must speak English

Exclusion Criteria:

* Patients under the age of 65

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population used will include all genders, socioeconomic, and ethnic backgrounds. Patients with (mild cognitive impairment, dementia) and without (normal cognition) a diagnosis of cognitive dysfunction will be included in the study. Geriatric patients (>65 years old) will be included in the study, but recruited caregivers must be over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Rapid Cognitive Screen Scores | 1 month
  Rapid Cognitive Screen scores with be done at home via telemedicine approximately 30 days after being done at a clinic visit. Scores range on a scale of 0-10. Scores will also be subdivided into the categories of free recall (5 points), clock drawing (4 points) and insight (1 point); and based on classification on the RCS (normal cognitive function, mild cognitive impairment [MCI], dementia).

SECONDARY OUTCOMES:
Clinical diagnosis of cognitive dysfunction (where available from medical records) will be compared to Rapid Cognitive Screen scores done at home via telemedicine | Previous clinical diagnosis cognitive dysfunction documented in medical records up to 36 months prior to Rapid Cognitive Screen scores done at home via telemedicine
  Diagnosis of mild cognitive impairment or dementia in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Theodore K Malmstrom, PhD, Principal Investigator — Saint Louis Univeristy
Locations (1):
- Saint Louis University Geriatric Clinic, St Louis, Missouri, United States

REFERENCES:
- [Background] van der Linde RM, Dening T, Stephan BC, Prina AM, Evans E, Brayne C. Longitudinal course of behavioural and psychological symptoms of dementia: systematic review. Br J Psychiatry. 2016 Nov;209(5):366-377. doi: 10.1192/bjp.bp.114.148403. Epub 2016 Aug 4. PMID 27491532
- [Background] Cordell CB, Borson S, Boustani M, Chodosh J, Reuben D, Verghese J, Thies W, Fried LB; Medicare Detection of Cognitive Impairment Workgroup. Alzheimer's Association recommendations for operationalizing the detection of cognitive impairment during the Medicare Annual Wellness Visit in a primary care setting. Alzheimers Dement. 2013 Mar;9(2):141-50. doi: 10.1016/j.jalz.2012.09.011. Epub 2012 Dec 20. PMID 23265826
- [Background] Malmstrom TK, Voss VB, Cruz-Oliver DM, Cummings-Vaughn LA, Tumosa N, Grossberg GT, Morley JE. The Rapid Cognitive Screen (RCS): A Point-of-Care Screening for Dementia and Mild Cognitive Impairment. J Nutr Health Aging. 2015 Aug;19(7):741-4. doi: 10.1007/s12603-015-0564-2. PMID 26193857
- [Background] Dubois B, Padovani A, Scheltens P, Rossi A, Dell'Agnello G. Timely Diagnosis for Alzheimer's Disease: A Literature Review on Benefits and Challenges. J Alzheimers Dis. 2016;49(3):617-31. doi: 10.3233/JAD-150692. PMID 26484931
- [Background] Weimer DL, Sager MA. Early identification and treatment of Alzheimer's disease: social and fiscal outcomes. Alzheimers Dement. 2009 May;5(3):215-26. doi: 10.1016/j.jalz.2009.01.028. Epub 2009 Apr 11. PMID 19362885
- [Background] Lin JS, O'Connor E, Rossom RC, Perdue LA, Eckstrom E. Screening for cognitive impairment in older adults: A systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2013 Nov 5;159(9):601-12. doi: 10.7326/0003-4819-159-9-201311050-00730. PMID 24145578

DOCUMENTS (1):
  • Study Protocol: EpxCogScreen (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03569722/Prot_000.pdf